CLINICAL TRIAL: NCT00376779
Title: A Phase II, Observer-blind, Randomized Study to Evaluate the Immunogenicity, Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Combined DssiTgdPa-HBV-IPV/Hib Vaccine Containing Diphtheria Toxoid From the Statens Serum Institute (SSI) of Denmark and Tetanus Toxoid From GSK Biologicals' Kft [GD], Compared to the Currently Licensed GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine (Infanrix Hexa TM) When Administered to Healthy Infants at 2, 3 and 4 Months of Age.
Brief Title: Immunogenicity and Safety of a DTPa-HBV-IPV/Hib Vaccine Given at 2, 3 and 4 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106786
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type b
Keywords: Haemophilus influenzae type b; Double-blind; Finland; randomized; phase 2; GSK Biologicals; DTPa-HBV-IPV/Hib
MeSH Terms: conditions — Tetanus; Diphtheria; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

INTERVENTIONS:
Biological: Infanrix hexa Vaccine

SUMMARY:
The purpose of this study is to show that the immunogenicity of newly formulated DTPa-HBV-IPV/Hib vaccine is as good as the immunogenicity of the currently licensed formulation of the vaccine. The vaccine will be administered as a primary vaccination course to healthy infants at 2, 3 and 4 months of age and its safety and reactogenicity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between, and including, 8 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parents/guardians of the subject.
* Born after a normal gestation period of 36 to 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs from birth until first primary vaccination dose.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration/planned administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the first dose and ending 30 days after the last dose, with the exception of the human rotavirus (HRV) vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B and/or Haemophilus influenza type b (Hib) vaccination or disease.
* Hepatitis B virus (HBV) vaccination at birth.
* History of seizures or progressive neurological disease.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Antibody concentration/response to all vaccine antigens after vaccination

SECONDARY OUTCOMES:
Solicited (D0-3); unsolicited events (D0-30); serious adverse events (SAEs) (full study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Finland (6):
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106786 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register